CLINICAL TRIAL: NCT04721067
Title: Treating Insomnia to Reduce Inflammation in HIV
Brief Title: HIV-related Insomnia and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Samir K. Gupta, MD, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21MH127206-01 (NIH); 1R21MH127206-01 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hiv; Insomnia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Initiation and Maintenance Disorders | interventions — Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study outcomes will be analyzed and compared by blinded investigators and statisticians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CBT-I (Experimental): This arm will receive internet CBT-I using SHUTi, a validated and proven therapy provided via internet in the general population.
  Interventions: Device: SHUTi
- Sleep Education/Hygiene (Active Comparator): This arm will receive best practices education on sleep hygiene.
  Interventions: Behavioral: Sleep Education/Hygiene

INTERVENTIONS:
Device: SHUTi — SHUTi is the empirically supported, internet CBT-I that is fully accessible via tablets and smartphones. It uses a self-guided, fully automated, interactive, multimedia format to deliver six 45-minute sessions, the structure and content of which mirror traditional face-to-face CBT-I. Session content includes sleep restriction, stimulus control, sleep hygiene, cognitive restructuring, and relapse prevention. SHUTi is enhanced through a variety of interactive features, including personalized goal setting, graphical feedback based on inputted symptoms, animations and illustrations to enhance comprehension, quizzes to test user knowledge, patient vignettes, and video-based expert explanation. Across sessions, patients also receive tailored sleep recommendations and feedback based on the sleep diary data they enter into the program.
  Arms: CBT-I
Behavioral: Sleep Education/Hygiene — A research assistant (RA) will deliver the active control procedures. During the first 4 weeks, the RA will have two calls with each control participant - one 45-minute call on insomnia education (including their HIV provider's role in its management) and one 45-minute call on sleep hygiene practices. To end the first call, the RA will email or mail a list of local behavioral health services to patients and will encourage them to follow-up with their HIV provider. We will then notify the HIV provider, which will encourage them to address their patient's insomnia and provide the same list of local services.
  Arms: Sleep Education/Hygiene

SUMMARY:
This randomized trial will determine the effects of internet cognitive behavioral therapy on measures of systemic inflammation in HIV-positive people receiving antiretroviral therapy.

DETAILED DESCRIPTION:
The primary objective of this pilot trial is to evaluate the effects of cognitive behavioral therapy for insomnia (CBT-I) on changes in circulating levels of hsCRP at 24 weeks in virologically-suppressed, HIV-positive adults with insomnia, defined as having an Insomnia Severity Index (ISI) score ≥ 11. Secondary objectives include comparing changes in hsCRP at 12 weeks, changes in other circulating inflammation biomarkers (IL-6, sCD14, sCD163, CD14+CD16+ monocytes) at both 12 and 24 weeks, and ISI scores and other self-reported patient outcomes at both 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented as listed clinically in the participant's electronic medical record by any of the following tests: (1) any licensed rapid HIV test, (2) HIV enzyme test kit at any time prior to study entry, (3) at least one detectable HIV-1 antigen, or (4) at least one detectable plasma HIV-1 RNA viral load.
* Age equal to or greater than 18 years.
* Ongoing receipt of stable antiretroviral therapy of any kind for at least 180 days prior to the date of the HIV-1 RNA value determining eligibility.
* HIV-1 RNA level < 75 copies/mL at Screening.

NOTE: There are no CD4 cell count eligibility criteria for this trial.

-ISI score ≥ 11 at Screening.

NOTE: Use of sleeping aids/medications is permitted as long as the ISI score criterion is met.

Exclusion Criteria:

* Inability to complete written, informed consent.
* Incarceration at the time of any study visit.
* Active suicidality at Entry, as determined by the patient's HIV provider or social worker following a positive response (1, 2, or 3) to PHQ-9 Item #9 and a positive response (yes) to one or more of the three questions (for Question #3, the previous attempt must be within the past 10 years) on the Patient Suicidality Form (see Appendix).
* Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosus, inflammatory bowel diseases, or other collagen vascular diseases).

NOTE: Hepatitis B or C co-infections are NOT exclusionary, but treatment for hepatitis C cannot be provided during study participation.

* End stage renal disease requiring renal replacement therapy (dialysis, transplantation).
* Known or suspected malignancy requiring systemic treatment within 180 days of the Entry Visit.

NOTE: Localized treatment for skin cancers is not exclusionary.

-Therapy for serious medical illnesses within 14 days prior to the Entry Visit.

NOTE: Therapy for serious medical illnesses that overlaps with a study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Pregnancy or breastfeeding during the course of the study.
* Receipt of investigational agents, cytotoxic chemotherapy, systemic immunosuppressive therapies, systemic glucocorticoids (of any dose), or anabolic steroids at the Entry Visit.

NOTE: Physiologic testosterone replacement therapy or topical steroids is not exclusionary. Inhaled/nasal steroids are not exclusionary as long as the participant is not also receiving HIV protease inhibitors.

* Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* History of bipolar disorder or a psychotic disorder, including schizophrenia.

NOTE: Depressive disorders are not exclusionary.

* Current sleep disorder diagnosis other than insomnia disorder (e.g., sleep apnea).
* Have a schedule requiring a bedtime earlier than 8:00pm or later than 2:00am or arising time earlier than 4:00am or later than 10:00am (thus preventing adoption of SHUTi interventions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Infectious Diseases Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We will fully participate in sharing our unique datasets and associated stored samples with other interested parties once the primary analyses have been completed. This dataset will include individual-level baseline, interim visit, ancillary, procedural-based, and outcome data. Data from scored assessments (e.g., psychosocial questionnaires) will include both raw data elements (e.g., individual item responses) and summary information (e.g., total scores) where feasible. Laboratory results will also be available as individual-level results from each study visit.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will become available once the primary results are analyzed and published.
Access Criteria: Data and sample requests will be honored after submission of a short proposal that outlines an important scientific question with an appropriate statistical analysis plan that justifies the use of these datasets. In addition, the requests must also verify that confidentiality of the datasets will be ensured.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT-I | Sleep Education/Hygiene
Started | 16 | 14
Completed | 12 | 10
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Sleep Education/Hygiene | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.9) | 52.6 (9.2) | 50.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 6 | 5 | 11
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Insomnia Severity Index (ISI) Score [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) total score will be measured. The total scale has a minimum score of 0 and a maximum score of 28, with higher scores indicating a worse outcome.
  units on a scale | 18.9 (6.0) | 16.6 (4.6) | 17.9 (5.4)
High Sensitivity C-Reactive Protein [Mean (Standard Deviation); unit: mg/L] | 4.3 (4.8) | 5.2 (6.4) | 4.7 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in hsCRP Levels at 24 Weeks
Description: Circulating high sensitivity C-reactive protein levels will be measured
Time Frame: Baseline and 24 weeks
Population: 12 and 9 participants, respectively, in the CBT-I and Sleep Education/Hygiene arms had hsCRP data collected at Week 24. The changes in hsCRP values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 12 | 9
mg/L | 2.19 (4.56) | 4.47 (20.12)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.607, Regression, Logistic; Adjusted for baseline values; Mean Difference (Net) = -2.27, 95% CI 2-sided [-15.14 to 10.60]

2. Secondary Outcome: Change in IL-6 Levels at 24 Weeks
Description: Circulating interleukin-6 levels will be measured. Interleukin-6 is a measure of systemic inflammation.
Time Frame: Baseline and 24 weeks
Population: The changes in IL-6 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 11
pg/mL | 0.66 (1.25) | 3.11 (11.03)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.766, ANCOVA; Mean Difference (Net) = -2.99, 95% CI 2-sided [-10.74 to 4.76]

3. Secondary Outcome: Change is sCD14 Levels at 24 Weeks
Description: Circulating soluble CD14 levels will be measured. Soluble CD14 is a measure of monocyte activation.
Time Frame: Baseline and 24 weeks
Population: The changes in sCD14 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 11
ng/mL | 1.37 (402.36) | -112.10 (500.22)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.465, ANCOVA; Mean Difference (Net) = 145.54, 95% CI 2-sided [-264.05 to 555.14]

4. Secondary Outcome: Change in sCD163 Levels at 24 Weeks
Description: Circulating soluble CD163 levels will be measured. Soluble CD163 is a measure of monocyte/macrophage activation.
Time Frame: Baseline and 24 weeks
Population: The changes in sCD163 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 11
ng/mL | 44.40 (212.58) | -89.37 (208.93)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.178, ANCOVA; Mean Difference (Net) = 137.79, 95% CI 2-sided [-68.71 to 344.30]

5. Secondary Outcome: Change in CD14+CD16+ Monocytes at 24 Weeks
Description: Circulating intermediate monocytes as defined by flow cytometric evaluation for CD14+CD16+ monocytes will be measured. CD14+CD16+ monocytes are measured by flow cytometry and indicate the pro-inflammatory subpopulation of monocytes.
Time Frame: Baseline and 24 weeks
Population: The changes in CD14+CD16+ monocyte values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: percentage of total monocytes
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 9
percentage of total monocytes | -0.30 (13.95) | 0.39 (3.13)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.548, ANCOVA; Mean Difference (Net) = 1.87, 95% CI 2-sided [-4.58 to 8.31]

6. Secondary Outcome: Change in hsCRP Levels at 12 Weeks
Description: Circulating high sensitivity C-reactive protein (hsCRP) levels will be measured. hsCRP is a measure of systemic inflammation.
Time Frame: Baseline and 12 weeks
Population: The changes in hsCRP values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
mg/L | 0.31 (1.86) | 0.85 (3.29)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.579, ANCOVA; Mean Difference (Net) = -0.67, 95% CI 2-sided [-3.14 to 1.80]

7. Secondary Outcome: Change in Insomnia Severity Index (ISI) at 24 Weeks
Description: The Insomnia Severity Index (ISI) total score will be measured. The total scale has a minimum score of 0 and a maximum score of 28, with higher scores indicating a worse outcome.
Time Frame: Baseline and 24 weeks
Population: The changes in ISI values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -7.48 (8.10) | -6.00 (3.59)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.766, ANCOVA; Mean Difference (Net) = -0.63, 95% CI 2-sided [-5.00 to 3.74]

8. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) at 24 Weeks
Description: Changes in the Pittsburgh Sleep Quality Index (PSQI) questionnaire global scores will be measured. The global PSQI score has a range from 0 to 21, with higher numbers indicating worse sleep quality.
Time Frame: Baseline and 24 weeks
Population: The changes in PSQI values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -3.40 (3.92) | -2.17 (3.33)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.42, ANCOVA; Mean Difference (Net) = -1.23, 95% CI 2-sided [-4.39 to 1.93]

9. Secondary Outcome: Change in Dysfunctional Beliefs and Attitudes About Sleep (DBAS-16) at 24 Weeks
Description: The Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) questionnaire total scores will be measured. The DBAS-16 total score ranges from 0 to 10, with higher scores indicating more dysfunctional beliefs and attitudes about sleep.
Time Frame: Baseline and 24 weeks
Population: The changes in DBAS-16 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -2.16 (1.45) | -1.96 (1.47)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.91, ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-1.34 to 1.20]

10. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) at 24 Weeks
Description: Patient Health Questionnaire (PHQ-9) scores will be measured. The PHQ-9 ranges from 0 to 27, with higher scores indicating worse depression symptom severity.
Time Frame: Baseline and 24 weeks
Population: The changes in PHQ-9 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -5.64 (7.68) | -4.27 (4.94)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.73, ANCOVA; Mean Difference (Net) = 0.79, 95% CI 2-sided [-4.03 to 5.60]

11. Secondary Outcome: Change in Hopkins Symptom Checklist (SCL-20) at 24 Weeks
Description: The Hopkins Symptom Checklist (SCL-20) questionnaire score will be measured. The SCL-20 questionnaire scores range from 0 to 4, where higher scores indicate more severe depressive symptoms.
Time Frame: Baseline and 24 weeks
Population: The changes in SCl-20 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -0.61 (0.75) | -0.64 (0.66)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.42, ANCOVA; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.30 to 0.68]

12. Secondary Outcome: Change in Generalized Anxiety Disorder-7 (GAD-7) at 24 Weeks
Description: The Generalized Anxiety Disorder-7 (GAD-7) questionnaire total score will be measured. The GAD-7 total score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Time Frame: Baseline and 24 weeks
Population: The changes in GAD-7 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | -3.08 (4.11) | -4.29 (4.01)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.18, ANCOVA; Mean Difference (Net) = 1.79, 95% CI 2-sided [-0.90 to 4.48]

13. Secondary Outcome: Change in PROMIS FACIT-F Fatigue Short Form at 24 Weeks
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) subscale questionnaire score ranges from 0 to 52, with higher scores indicating greater fatigue.
Time Frame: Baseline and 24 weeks
Population: The changes in PROMIS FACIT-F values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | 3.21 (10.28) | 1.36 (5.85)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.48, ANCOVA; Mean Difference (Net) = -2.03, 95% CI 2-sided [-7.97 to 3.90]

14. Secondary Outcome: Change in Alcohol Use Disorders Identification Test (AUDIT) at 24 Weeks
Description: Alcohol Use Disorders Identification Test (AUDIT) questionnaire total scores will be measured. The AUDIT total score ranges from 0 to 40, with higher scores indicating greater likelihood of alcohol dependence.
Time Frame: Baseline and 24 weeks
Population: The changes in AUDIT values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 9 | 11
score on a scale | -0.22 (1.72) | -2.36 (3.64)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.08, ANCOVA; Mean Difference (Net) = 1.42, 95% CI 2-sided [-0.24 to 3.08]

15. Secondary Outcome: Change in Short Form-36 (SF-36) Health Survey and 24 Weeks
Description: Short Form-36 (SF-36) general health total questionnaire scores will be measured. The SF-36 general health total score ranges from 0 to 100, with higher scores indicating better general health.
Time Frame: Baseline and 24 weeks
Population: The changes in SF-36 values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
score on a scale | 7.50 (18.45) | 7.29 (11.45)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.94, ANCOVA; Mean Difference (Net) = 0.51, 95% CI 2-sided [-13.50 to 14.52]

16. Secondary Outcome: Use of Sleep Medications at Week 12
Description: The number of sleep medications used by each participant at Week 12
Time Frame: Week 12
Population: This measure was mistakenly not collected by the study team and is considered a protocol deviation.
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Use of Sleep Medications at Week 24
Description: The number of sleep medications used by each participant at Week 24
Time Frame: Week 24
Population: This measure was mistakenly not collected by the study team and is considered a protocol deviation.
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Insomnia Treatment Satisfaction at Week 12
Description: An assessment of the participant's satisfaction with their assigned insomnia treatment at Week 12, ranging from 1-5, with lower scores indicating greater overall treatment satisfaction.
Time Frame: Week 12
Population: The changes in insomnia treatment satisfaction values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 12
units on a scale | 3.10 (0.74) | 2.67 (1.15)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.45 to 1.32]

19. Secondary Outcome: Insomnia Treatment Satisfaction at Week 24
Description: An assessment of the participant's satisfaction with their assigned insomnia treatment at Week 24, ranging from 1-5, with lower scores indicating greater overall treatment satisfaction.
Time Frame: Week 24
Population: The changes in insomnia treatment satisfactin values are only reported for those who had paired values at Baseline and Week 24 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 9 | 12
units on a scale | 3.00 (0.87) | 2.75 (1.22)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.75 to 1.25]

20. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) at 12 Weeks
Description: as for outcome 8
Time Frame: Baseline and 12 weeks
Population: The changes in PSQI values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 11
score on a scale | -3.00 (4.11) | -1.91 (3.21)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.52, ANCOVA; Mean Difference (Net) = -1.05, 95% CI 2-sided [-4.42 to 2.31]

21. Secondary Outcome: Change in Dysfunctional Beliefs and Attitudes About Sleep (DBAS-16) at 12 Weeks
Description: as for outcome 9
Time Frame: Baseline and 12 weeks
Population: The changes in DBAS-16 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -2.07 (2.52) | -1.47 (1.58)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.61, ANCOVA; Mean Difference (Net) = -0.44, 95% CI 2-sided [-2.20 to 1.32]

22. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) at 12 Weeks
Description: as for outcome 10
Time Frame: Baseline and 12 weeks
Population: The changes in PHQ-9 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -1.82 (9.47) | -3.10 (4.25)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.16, ANCOVA; Mean Difference (Net) = 3.68, 95% CI 2-sided [-1.61 to 8.97]

23. Secondary Outcome: Change in Hopkins Symptom Checklist (SCL-20) at 12 Weeks
Description: as for outcome 11
Time Frame: Baseline and 12 weeks
Population: The changes in SCL-20 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -0.37 (1.01) | -0.59 (0.60)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.13, ANCOVA; Mean Difference (Net) = 0.43, 95% CI 2-sided [-0.13 to 1.00]

24. Secondary Outcome: Change in Generalized Anxiety Disorder-7 (GAD-7) at 12 Weeks
Description: as for outcome 12
Time Frame: Baseline and 12 weeks
Population: The changes in GAD-7 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -0.71 (5.16) | -3.88 (5.32)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.03, ANCOVA; Mean Difference (Net) = 3.88, 95% CI 2-sided [0.35 to 7.41]

25. Secondary Outcome: Change in PROMIS FACIT-F Fatigue Short Form at 12 Weeks
Description: as for outcome 13
Time Frame: Baseline and 12 weeks
Population: The changes in PROMIS FACIT-F values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -0.02 (12.16) | 0.72 (5.38)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.41, ANCOVA; Mean Difference (Net) = -3.20, 95% CI 2-sided [-11.07 to 4.66]

26. Secondary Outcome: Change in Alcohol Use Disorders Identification Test (AUDIT) at 12 Weeks
Description: as for outcome 14
Time Frame: Baseline and 12 weeks
Population: The changes in AUDIT values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 10 | 10
score on a scale | 0.70 (3.27) | -1.00 (1.70)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.17, ANCOVA; Mean Difference (Net) = 1.70, 95% CI 2-sided [-0.83 to 4.22]

27. Secondary Outcome: Change in Short Form-36 (SF-36) Health Survey and 12 Weeks
Description: as for outcome 15
Time Frame: Baseline and 12 weeks
Population: The changes in SFl-36 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | 10.45 (17.24) | 7.19 (11.31)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.58, ANCOVA; Mean Difference (Net) = 3.49, 95% CI 2-sided [-9.58 to 16.55]

28. Secondary Outcome: Change in IL-6 Levels at 12 Weeks
Description: Circulating interleukin-6 levels will be measured. Interleukin-6 is a measure of systemic inflammation.
Time Frame: Baseline and 12 weeks
Population: The changes in IL-6 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
pg/mL | 0.05 (0.64) | 1.24 (3.99)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.74, ANCOVA; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.79 to 1.10]

29. Secondary Outcome: Change is sCD14 Levels at 12 Weeks
Description: Circulating soluble CD14 levels will be measured. Soluble CD14 is a measure of monocyte activation.
Time Frame: Baseline and 12 weeks
Population: The changes in sCD14 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
ng/mL | 57.43 (276.42) | -63.31 (149.77)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.17, ANCOVA; Mean Difference (Net) = 129.077, 95% CI 2-sided [-57.78 to 315.92]

30. Secondary Outcome: Change in sCD163 Levels at 12 Weeks
Description: Circulating soluble CD163 levels will be measured. Soluble CD163 is a measure of monocyte/macrophage activation.
Time Frame: Baseline and 12 weeks
Population: The changes in sCD163 values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
ng/mL | 95.00 (309.05) | 22.51 (143.62)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.31, ANCOVA; Mean Difference (Net) = 109.71, 95% CI 2-sided [-108.37 to 327.78]

31. Secondary Outcome: Change in CD14+CD16+ Monocytes at 12 Weeks
Description: as for outcome 5
Time Frame: Baseline and 12 weeks
Population: The changes in CD14+16+ monocyte values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: percentage of total monocytes
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 9 | 11
percentage of total monocytes | -1.75 (9.83) | 0.23 (3.62)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.92, ANCOVA; Mean Difference (Net) = 0.24, 95% CI 2-sided [-4.52 to 5.00]

32. Secondary Outcome: Change in Insomnia Severity Index (ISI) at 12 Weeks
Description: as for outcome 7
Time Frame: Baseline and 12 weeks
Population: The changes in ISI values are only reported for those who had paired values at Baseline and Week 12 to assess change in this variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Education/Hygiene
Number analyzed (Participants) | 11 | 12
score on a scale | -5.67 (8.62) | -3.92 (5.07)
Statistical Analysis 1: Comparison: CBT-I vs Sleep Education/Hygiene; Test type: Superiority; p = 0.66, ANCOVA; Mean Difference (Net) = -1.11, 95% CI 2-sided [-6.28 to 4.06]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | CBT-I | Sleep Education/Hygiene
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04721067/Prot_006.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04721067/SAP_011.pdf
  • Informed Consent Form (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04721067/ICF_008.pdf